CLINICAL TRIAL: NCT03290586
Title: Fusion Rates and Cost Analysis of Patients Undergoing 1st Metatarsal Phalangeal Joint Arthrodesis; the Evaluation of a Novel, Single Use Sterile, Disposable Delivery System
Brief Title: Fusion Rates and Cost Analysis of Patients Undergoing 1st Metatarsal Phalangeal Joint Arthrodesis
Status: Completed | Type: Observational
Sponsor: JEM Research Institute (Industry)
Collaborators: Flower Orthopedics (Unknown)
Responsible Party: Principal Investigator, John Levin, Principal Investigator, JEM Research Institute
Other Study IDs: FLO-001
Record Dates: First submitted 2017-09-18; First posted 2017-09-25 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: First Metatarsophalangeal Joint Arthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Flower Cube — single use, sterile disposable fixation construct

SUMMARY:
This is a longitudinal, multi-center study to be conducted in at least five institutions from the private surgeon offices. These surgeons will collect data from X-rays, wound complications \and hardware complications.

ELIGIBILITY:
Inclusion Criteria:

* Painful Hallux Limitus or Rigidus
* Painful Geriatric Hallux Valgus
* Failed prior 1st MTP joint arthroplasty (hemi-total)
* Arthritis of any etiology other than degenerative causes

Exclusion Criteria:

* Age less than 18 years
* Pregnant Females
* Active or prior infection at the target joint
* Immunocompromised patients
* Patients unwilling to sign informed consent
* Patient's unwilling to participate the in study protocol
* Subject with known sensitivity to titanium implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the surgeons' private practices. These patients have already met the criteria for surgical intervention and have agreed to undergo the operative procedure and postoperative management.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

PRIMARY OUTCOMES:
Union Rates | 12 months
  Confirm union rates comparable to existing outcomes complications with our proposed construct.
Hardware Failures | 12 months
  Evaluate hardware failures with our proposed construct.
Complications | 12 months
  Evaluate complications with the procedure

SECONDARY OUTCOMES:
Cost Data | 12 months
  Review cost data using the Flower Orthopedics single use, sterile disposable fixation construct performed in an outpatient surgical setting compared to in patient hospital setting.

CONTACTS AND LOCATIONS:
Overall Officials: John Levin, DPM, Principal Investigator — JEM Research Institute
Locations (1):
- JEM Research Institute, Atlantis, Florida, United States

IPD SHARING:
Plan to Share IPD: No